CLINICAL TRIAL: NCT00627380
Title: Yoga for the Management of HIV-Metabolic Syndromes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Kevin E. Yarasheski/Principal Investigator, Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT003083 (NIH); R21AT003083 (NIH); WU187
Record Dates: First submitted 2008-02-28; First posted 2008-03-03 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: HIV Infections; HIV Metabolic Cardiovascular Syndrome; HIV Lipodystrophy; HIV Metabolic Syndromes; Hypertension
Keywords: HIV; AIDS; insulin resistance; diabetes; dyslipidemia; visceral adiposity; subcutaneous adipose wasting; cardiovascular disease; hypertension; endothelial function; quality of life; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Hypertension; Acquired Immunodeficiency Syndrome; Insulin Resistance; Diabetes Mellitus; Dyslipidemias; Cardiovascular Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STOC (Placebo Comparator): Standard of care arm continues to receive standard of care treatment for HIV, but does not receive any new treatment/intervention or change in anti-HIV medications. Runs parallel to experimental group. At the end of this 16-wk control period, participants are invited to crossover into the experimental group
  Interventions: Other: Standard of care
- YOGA (Experimental): Yoga lifestyle intervention administered by certified yoga instructor.
  Interventions: Behavioral: Yoga lifestyle intervention

INTERVENTIONS:
Behavioral: Yoga lifestyle intervention — Sixteen weeks of 2-3 yoga sessions per week, 1.5 hrs per session administered by a certified yoga instructor. Sessions include breathing exercises and yoga postures/positions.
  Other Names: Hatha yoga; Ashtanga yoga
  Arms: YOGA
Other: Standard of care — Participants are observed/followed for 16 weeks during which lifestyle and medication changes are discouraged, unless medically necessary.
  Other Names: Observation control group
  Arms: STOC

SUMMARY:
We are testing the safety and efficacy of a 16-wk yoga lifestyle intervention on oral glucose tolerance, fasting lipid/lipoprotein levels, body composition, cardiovascular function, quality of life, CD4+ T-cell counts and viral load in HIV-infected men and women with components of The Metabolic Syndrome. We hypothesize that a yoga lifestyle intervention will improve metabolic, anthropometric, cardiovascular disease parameters, and quality of life domains without adversely affecting immune or virologic status in people living with HIV.

DETAILED DESCRIPTION:
Very few safe, effective, and novel treatments for metabolic syndromes that develop in HIV-infected people exist. These metabolic syndromes may increase cardiovascular disease risk in HIV-infected people and may reduce their quantity and quality of life. Practicing a yoga lifestyle intervention may provide a safe, effective and novel therapy for HIV metabolic syndromes, but this alternative form of therapy has not been tested in HIV-infected people with metabolic syndromes. In men and women with HIV-related metabolic syndromes, we will determine:

1. The safety of practicing a yoga lifestyle in HIV-infected people treated with HAART who are experiencing metabolic and anthropometric syndromes.
2. To quantify the effects of practicing a yoga lifestyle on metabolic and anthropomorphic syndromes in HIV-infected people treated with HAART who are experiencing these syndromes.
3. To quantify the effects of practicing a yoga lifestyle on cardiovascular disease (CVD) risk in HIV-infected people treated with HAART who are at increased CVD risk because of existing metabolic and anthropomorphic syndromes.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected volunteers must have dyslipidemia (fasting serum LDL-cholesterol >100mg/dL, or
* triglycerides >200mg/dL, or
* HDL-cholesterol <40mg/dL (men) or <50mg/dL (women), or
* impaired glucose tolerance (fasting blood glucose 100-140mg/dL or
* fasting insulin 13-45µU/mL or 2hr glucose during the oGTT 140-200mg/dL),or
* central adiposity (waist circumference >102 cm (40inches in men) or >88cm (35inches in women)
* The purpose is to identify and enroll participants with a clear proatherogenic lipid profile
* increased CVD risk
* abdominal adiposity, and fasting glucose intolerance or insulin resistance
* but not type 2 diabetics who have normalized their blood sugars using glucose-lowering agents. If a type 2 diabetic uses a glucose-lowering medication, but they are still insulin resistant/glucose intolerant (by above criteria), they are eligible to participate, because we are testing the added benefits of yoga therapy on a defined dysmetabolic syndrome in participants who are stable on the standard-of-care for these metabolic syndromes, and this includes glucose- and lipid-lowering agents
* These criteria must be met, even in volunteers receiving glucose- or lipid-lowering agents, so that we enroll participants who have developed metabolic syndromes that are not normalized by traditional pharmacologic approaches
* Volunteers receiving glucose- or lipid-lowering agents who have normalized their lipid, glucose and insulin levels below these defined limits, are not eligible to enroll.

Additional Inclusion Criteria.

* 18-70 years old.
* Plasma HIV RNA <15,000 copies/ml for previous 3months.
* CD4 count >200 c/µL for previous 3 months.
* Stable HIV RNA level and stable CD4 count for at least the past 3 months. Some HIV-infected people can accomplish this while not receiving HAART (eg. long term non-progressors) and will be included. But, most of the participants will be on a HAART regimen that includes either 2 NRTIs + NNRTI, or 2NRTIs + PI, or NRTI+NNRTI+PI
* "Normal" blood chemistries for at least 1 month prior to enrollment:

  * platelet count >30,000/mm3
  * absolute neutrophil count >750/mm3
  * transaminases <5x the upper limit of normal
  * creatinine <3x the upper limit of normal
  * albumin >30g/L

Exclusion Criteria:

* Chronic hepatitis B infection (HB surface antigen positive). Active hepatitis C infection (detectable Hep C RNA). Those who have cleared hepatitis B or C infection are eligible.
* Diabetes [fasting glucose >140 mg/dL, or fasting insulin >45 µU/mL, or 2-hr glucose >200mg/dL].
* History of diabetes mellitus that pre-dates HIV-infection. Medications or agents that regulate glucose or lipid metabolism (e.g., insulin-sensitizers, insulin-secretagogues, HMG-CoA reductase inhibitors ('statins'), fibrates, niacin) are permitted. A large percentage of ACTU subjects and ID Clinic patients receiving RTV-boosted regimens are also receiving lipid-lowering agents. Excluding them might significantly reduce the pool of potential enrollees. The glucose- or lipid-lowering agent and dose must be stable for at least 3 months prior to screening. Additionally, volunteers taking glucose-or lipid-lowering agents must still have dyslipidemia and impaired glucose tolerance criteria (above). If they are taking these agents and have 'normalized' their lipids/lipoproteins and hyperinsulinemia, then they are not eligible
* Gestational diabetes, pregnancy, or nursing mothers. Menstruating women must have a negative urine pregnancy test within 14 days prior to DEXA testing (minor radiation exposure from DEXA). To control for potential metabolic effects of alterations in female hormones during the menstrual cycle, all menstruating women will be tested during the follicular phase.
* Hypogonadism [total testosterone <200ng/dL (men) or <15ng/dL (women)]; thyroid disorder [TSH <0.2 or >12µIU/mL]; hypercortisolemia [morning cortisol >22µg/dL]. Replacement testosterone or thyroid hormones or human growth hormone to normalize abnormal levels is acceptable, as long as treatment has been stable, and blood testosterone, TSH or IGF-1 levels are within the normal range.
* Unwilling or unable to attend supervised yoga sessions 3days/wk provided by Brentwood Center for Health at the Connectcare Clinic. Any condition that might be contraindicated for yoga therapy (disabling neuromuscular or musculoskeletal injury/disorder)
* History of serious cardiovascular disease; MI, unstable angina, heart failure, congenital heart disease, coronary artery disease, resting ST-segment depression >1mm, coronary artery bypass graft, stroke, sinus tachycardia, arrhythmias, premature atrial or ventricular contractions, claudication. Bundle branch block is exclusionary because it limits the interpretability of the resting/exercise ECG. Cardiovascular contraindications to maximal exercise testing
* Anticipated change in anti-HIV medications or other medications that affect metabolism, within the next 4months
* Well-trained athletes (defined as >3 exercise training exposures/week; >30min regimented exercise/exposure maintained for at least the prior 4 weeks)
* Active substance abuse (eg, alcoholism, cocaine, heroin, crack, methamphetamine, phencyclidine)
* Active secondary infection or a significant change in chronic suppressive therapy for an opportunistic infection during 1 month prior to enrollment
* New serious systemic infection during the 3 weeks prior to enrollment
* Recent episode of hyperlactatemia or lactic acidosis, esp. with rapid weight loss
* Chronic renal insufficiency/failure or other comorbid conditions (eg. cancer, COPD) that alter metabolism
* Pancreatitis, celiac disease, or cirrhosis
* Inadequate macronutrient or energy intake, or malabsorptive disorder as determined by the research dietician
* Dementia or any condition that would prevent voluntary informed consent or compliance
* Other compounds or blinded investigational new drugs that might affect metabolism or confound data interpretation (eg. RU486, interleukin therapy, or cytokine-receptor antagonist)
* Oral glucocorticoid or corticosteroid use within the previous 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome is a metabolic parameter: insulin integrated area under the curve (AUC) during the oral glucose tolerance test. | Baseline and week 16

SECONDARY OUTCOMES:
Fasting lipid/lipoprotein levels. | Baseline and week 16
Body composition: visceral and subcutaneous adipose tissue areas (VAT, SAT), trunk/limb adipose ratio. | Baseline and week 16
Cardiovascular disease risk: Framingham 10-yr CVD risk calculation | Baseline and week 16
Quality of life: SF36 MOS | Baseline and week 16
Safety: CD4 count and plasma HIV RNA | Baseline and week 16

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Yarasheski, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Innes KE, Vincent HK. The influence of yoga-based programs on risk profiles in adults with type 2 diabetes mellitus: a systematic review. Evid Based Complement Alternat Med. 2007 Dec;4(4):469-86. doi: 10.1093/ecam/nel103. PMID 18227915
- [Background] Schambelan M, Wilson PW, Yarasheski KE, Cade WT, Davila-Roman VG, D'Agostino RB Sr, Helmy TA, Law M, Mondy KE, Nachman S, Peterson LR, Worm SW; Working Group 5. Development of appropriate coronary heart disease risk prediction models in HIV-infected patients. Circulation. 2008 Jul 8;118(2):e48-53. doi: 10.1161/CIRCULATIONAHA.107.189627. Epub 2008 Jun 19. No abstract available. PMID 18566316
- [Background] Bashir A, Laciny E, Lassa-Claxton S, Yarasheski KE. Magnetic resonance imaging for quantifying regional adipose tissue in human immunodeficiency virus-infected persons with the cardiometabolic syndrome. J Cardiometab Syndr. 2008 Spring;3(2):115-8. doi: 10.1111/j.1559-4572.2008.07595.x. No abstract available. PMID 18453813
- [Background] Cade WT, Yarasheski KE. Cardiometabolic disease in the human immunodeficiency virus: the tip of the iceberg? J Cardiometab Syndr. 2008 Spring;3(2):77-8. doi: 10.1111/j.1559-4572.2008.07204.x. No abstract available. PMID 18453805
- [Background] Mondy KE, de las Fuentes L, Waggoner A, Onen NF, Bopp CS, Lassa-Claxton S, Powderly WG, Davila-Roman V, Yarasheski KE. Insulin resistance predicts endothelial dysfunction and cardiovascular risk in HIV-infected persons on long-term highly active antiretroviral therapy. AIDS. 2008 Apr 23;22(7):849-56. doi: 10.1097/QAD.0b013e3282f70694. PMID 18427203
- [Result] Mondy K, Cade WT, Reeds DN, Lassa-Claxton S, Bopp C, Tucker S, Yarasheski KE. Hatha/Ashtanga yoga intervention modestly improves cardiovascular disease (CVD) risk parameters in dyslipidemic HIV+ subjects with central adiposity(abstract). Antiviral Ther. 12 (suppl 2):L47, 2007.
- [Result] Cade WT, Reeds DN, Mondy KE, Overton ET, Grassino J, Tucker S, Bopp C, Laciny E, Hubert S, Lassa-Claxton S, Yarasheski KE. Yoga lifestyle intervention reduces blood pressure in HIV-infected adults with cardiovascular disease risk factors. HIV Med. 2010 Jul 1;11(6):379-88. doi: 10.1111/j.1468-1293.2009.00801.x. Epub 2010 Jan 5. PMID 20059570